CLINICAL TRIAL: NCT02857673
Title: A Medical Home-Based Intervention to Prevent Child Neglect in High-Risk Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-35533; R01CE002820-01 (NIH)
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Child Abuse
Keywords: Children with Special Health Care Needs; Violence Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive Child Abuse Prevention Problem Solving (CAPPS), a one-on-one, workbook-based intervention of six sessions, each lasting approximately 30-60 minutes. CAPPS is intended to be delivered over a period of 12 weeks, with sessions occurring every 1-2 weeks. Sessions will be delivered at the medical home by bachelor level providers, whose availability and level of training mimic those of existing medical home care coordinators.
  Interventions: Behavioral: Child Abuse Prevention Problem Solving
- Active Control Group (Active Comparator): Parents in both study groups will receive the standard medical and social work services offered in the patient-centered medical homes where their children receive care. In addition, to account for potential surveillance bias, families in the control group will be contacted by a member of the study team six times over 12 weeks, approximating the frequency of contact that the intervention group receives from the CAPPS providers. The study team member will not be trained in CAPPS and will adhere to a case management model consistent with resources available in the medical home, checking in with control families and offering to help identify existing clinic and community resources as needed.
  Interventions: Behavioral: Active Control Group

INTERVENTIONS:
Behavioral: Child Abuse Prevention Problem Solving — The CAPPS intervention includes problem solving, motivational interviewing, and referral to existing services. Intervention providers will conduct three core problem solving sessions and three sessions tailored to the common problems experienced by parents of CSHCN: caregiver burden, difficulties navigating complex medical services, and social isolation. Intervention providers will use their motivational interviewing skills during regular, ongoing interactions with their clients to enhance willingness to participate meaningfully in CAPPS sessions. Referral to existing services in the medical home and in the community will occur as needs arise during CAPPS sessions.
  Other Names: CAPPS
  Arms: Intervention Group
Behavioral: Active Control Group — Parents in both study groups will receive the standard medical and social work services offered in the patient-centered medical homes where their children receive care. In addition, to account for potential surveillance bias, families in the control group will be contacted by a member of the study team six times over 12 weeks, approximating the frequency of contact that the intervention group receives from the CAPPS providers.
  Arms: Active Control Group

SUMMARY:
Child maltreatment, particularly neglect, disproportionally affects low-income children with special health care needs (CSHCN) and has serious short and long-term consequences. Currently, few replicable, evidence-based preventive services exist for such families, particularly within the context of the patient-centered medical home. Child Abuse Prevention Problem Solving (CAPPS), a targeted problem solving intervention that addresses key risk and protective factors for child neglect, has the potential to improve key parenting skills and overall wellbeing, ultimately improving outcomes for high-risk children. This study is a multi-center randomized controlled efficacy trial of CAPPS to determine the impact on child neglect, adherence to recommended medical care, and family stressors and strengths.

DETAILED DESCRIPTION:
Child maltreatment, particularly neglect, disproportionally affects low-income CSHCN and has serious short and long-term consequences. Currently, few replicable, evidence-based preventive services exist for such families, particularly within the context of the patient-centered medical home. CAPPS, a targeted problem solving intervention that addresses key risk and protective factors for child neglect, has the potential to improve key parenting skills and overall wellbeing, ultimately improving outcomes for high-risk children.

This is a multi-center randomized controlled efficacy trial of Child Abuse Prevention Problem Solving (CAPPS), a targeted intervention designed to address specific stressors faced by low-income parents of children with special health care needs (CSHCN) and to enhance family strengths previously been shown to reduce the risk of maltreatment. The study will enroll 250 parents of CSHCN who receive primary care in a network of urban patient-centered medical homes. The specific research aims are to 1: Decrease referrals to child protective services for neglect and increase adherence to recommended medical care; and 2: Decrease perceived social isolation, difficulty navigating complex services, and caregiver burden and enhance family strengths, including parental resilience, social connections, access to support in times of need, and knowledge of parenting and child development.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child under age 7 with a physical, emotional, or behavioral health condition
* Child on Medicaid
* Fluent in English or Spanish

Exclusion Criteria:

* Prior history of substantiated child maltreatment
* Prior history of report to child protective services for suspected child maltreatment
* Parent cognitively limited

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Referral to Child Protective Services for neglect | Up to 12 months after enrollment in study
  This will be determined using chart review and parent report.
Adherence to recommended medical care | Up to 12 months after enrollment in study
  Adherence will be evaluated by chart review to determine a composite measure that includes numbers of medical visits attended, hospitalizations, missed appointments, delayed or missed prescriptions fills, and receiving recommended immunizations.

SECONDARY OUTCOMES:
Parental resilience and social connections - CHIP | Up to 12 months after enrollment in study
  The Coping Health Inventory for Parents (CHIP) is a valid and reliable 45-item instrument designed to measure parents' response to managing family life when they have an ill child. It comprises three subscales (family integration, α=0.79; psychological stability, α=0.79; and understanding the child's medical situation, α=0.71) within which total mean scores are calculated.
Parental resilience and social connections - PM | Up to 12 months after enrollment in study
  The Pearlin Mastery Scale (PM) measures the degree to which individuals perceive themselves as in control of their lives.
Parental resilience and social connections - RSES | Up to 12 months after enrollment in study
  Rosenberg Self-esteem Scale (RSES).
Parental resilience and social connections - PSS | Up to 12 months after enrollment in study
  Perceived Stress Scale (PSS) - Stress domains include unpredictability, lack of control, burden overload, and stressful circumstances. Reliability studies show Cronbach α's of 0.78 -0.86. The PSS correlates with inventories of burnout & somatization.
Parental resilience and social connections - PSI | Up to 12 months after enrollment in study
  Parenting Stress - Short Form (PSI) - The PSI assesses a wide range of parenting behaviors in a single instrument, including attachment to child, social isolation, competence, relationship with spouse, and parental health. Cronbach's α for the parent domain is 0.93 and the test-retest coefficient is 0.96.
Parental resilience and social connections - SAS-SR | Up to 12 months after enrollment in study
  Social Adjustment Scale Self-Report (SAS-SR) - We will use the SAS-SR, which examines social and role functioning in six areas: work; social activities; relationships with family; spouse or partner; parent; member of family unit. The SAS has high internal consistency (α=0.74) and test-retest reliability (r=0.80). It is sensitive to change in depressed patients undergoing treatment.
Parental resilience and social connections - MOS-SS | Up to 12 months after enrollment in study
  Medical Outcomes Survey Social Support (MOS-SS) - This tool comprises 4 functional support scales (emotional/informational, tangible, affectionate, and positive interaction) and an overall social support index. Subscales are reliable (α's > 0.91).
Access to concrete support | Up to 12 months after enrollment in study
  This will be measured using the WE-CARE survey. The survey consists of 14 questions used to identify seven unmet material needs (education, employment, food security, housing, childcare, household heat, language) and has been tested previously with low-income parents in the clinic setting.
Knowledge of parenting skills, child development - PS | Up to 12 months after enrollment in study
  Parenting Scale (PS) - The parenting scale is a 30-item questionnaire that measures parenting practices and consistency around discipline, with a focus on dysfunctional discipline: laxness, over-reactivity, and hostility. The scale has good internal consistency (α = 0.78-0.85) and test-retest reliability.
Knowledge of parenting skills, child development - CTSPC | Up to 12 months after enrollment in study
  Parent-Child Conflict Tactics Scale (CTSPC) - This measure contains 5 subscales that look at different types of discipline. The measure has been validated and is used extensively in the child maltreatment literature.

OTHER OUTCOMES:
Problem solving skills | Up to 12 months after enrollment in study
  Problem solving skills will be measured using the Social Problem Solving Inventory -Revised (SPSI-R). This 25 item instrument measures problem orientation and problem-solving skills in 5 dimensions: positive and negative orientation; avoidance; impulsivity; and rationality. The SPSI-R was validated with a diverse community sample and norms exist for adolescents and young adults. It is highly correlated with mood among caregivers of children with disabilities. Subscale internal consistency scores range from 0.76-0.92; test-retest reliability is reported in the range of 0.72-0.88.
Depression symptoms | Up to 12 months after enrollment in study
  We will measure caregiver depression using the Quick Inventory of Depressive Symptomatology (QIDS) - Because the QIDS has a wide scoring range, it can be used to detect depressive illness in populations with moderate and low-level symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline J Kistin, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No